CLINICAL TRIAL: NCT06480396
Title: An International, Partially-randomised, Patient-preference Trial Within a Registry of High Versus Lower Intensity Radiological Surveillance Following Primary Resection of Retroperitoneal, Abdominal and Pelvic Soft Tissue Sarcoma
Brief Title: High Versus Lower Intensity Surveillance Following Resection of Retroperitoneal Sarcoma
Acronym: SARveillance
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: University of Birmingham (Other); University Hospital Birmingham NHS Foundation Trust (Other); Royal Marsden NHS Foundation Trust (Other); University Hospital Padova (Other); Campus Bio-Medico University (Other); The Netherlands Cancer Institute (Other); KU Leuven (Other); Heidelberg University (Other); Dana-Farber/Brigham and Women's Cancer Center (Other); Emory University (Other); Mayo Clinic (Other); Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium (Other); The Cleveland Clinic (Other); M.D. Anderson Cancer Center (Other); University of Southern California (Other); Ohio State University (Other); Ottawa Hospital Research Institute (Other); McGill University (Other); Peter MacCallum Cancer Centre, Australia (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INT201/16(05/23)
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-06

CONDITIONS: Sarcoma,Soft Tissue; Sarcoma Retroperitoneal
Keywords: Surveillance; Radiology; Surgery; Quality of life; Cost-effectiveness
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: Patients that are willing to be randomised will be allocated in a 1:1 ratio to a high or lower intensity follow-up schedule. The trial design is partially randomised controlled and partly patient choice with patient preference arms (PPAs) for those that decline randomisation. Patients fulfilling the inclusion criteria and willing to be recruited will be stratified by tumour grade and then randomised to either high or lower intensity surveillance. Patients who decline randomisation will subsequently be offered the opportunity to participate within the PPAs. The PPAs will allow participating patients to choose either high or lower intensity surveillance arms. The data generated from the PPAs will not be included in the comparison of randomised arms. However, they will give important insight into patients' motivations in choosing high or lower intensity surveillance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-intensity radiological surveillance (Experimental): High/intermediate grade histology: 3-4 monthly CT scan up to 2-years postoperatively, 6-monthly CT scan from 2-5 years postoperatively (schedule 1)
  Low grade histology: 6-monthly CT scan up to 2-years postoperatively, annual CT scan from 2-5 years postoperatively (schedule 2)
  Interventions: Diagnostic Test: High-intensity radiological surveillance
- Lower-intensity radiological surveillance (Active Comparator): High intermediate grade histology: 6-monthly CT scan up to 2-years postoperatively, annual CT scan from 2-5 years postoperatively (schedule 2)
  Low grade histology: Annual CT scan up to 2-years postoperatively, 18 monthly CT scan from 2-5 years postoperatively (schedule 3)
  Interventions: Diagnostic Test: Lower-intensity radiological surveillance

INTERVENTIONS:
Diagnostic Test: High-intensity radiological surveillance — The standard approach to surveillance imaging will be contrasted CT (IV and oral contrast) of the chest, abdomen and pelvis. All patients require radiological assessment of the chest, abdomen and pelvis at each surveillance round. Tolerance will be given in the protocol for selected patients where CT is not suitable to receive alternative imaging such as MRI or combination of MRI and CT. Uncontrasted CT imaging is permissible where renal toxicity or allergy from intravenous contrast is of concern. The use of plain radiography is not permitted as an alternative to CT imaging of the chest.
  Arms: High-intensity radiological surveillance
Diagnostic Test: Lower-intensity radiological surveillance — The standard approach to surveillance imaging will be contrasted CT (IV and oral contrast) of the chest, abdomen and pelvis. All patients require radiological assessment of the chest, abdomen and pelvis at each surveillance round. Tolerance will be given in the protocol for selected patients where CT is not suitable to receive alternative imaging such as MRI or combination of MRI and CT. Uncontrasted CT imaging is permissible where renal toxicity or allergy from intravenous contrast is of concern. The use of plain radiography is not permitted as an alternative to CT imaging of the chest.
  Arms: Lower-intensity radiological surveillance

SUMMARY:
The SARveillance trial is an efficient, pragmatic, multi-centre, international, stratified, partially-randomised, patient-preference trial within a registry of high versus lower intensity radiological surveillance following primary resection of retroperitoneal, abdominal and pelvic soft tissue sarcoma. The trial design is stratified by sarcoma tumour grade (high/intermediate grade and low grade).

DETAILED DESCRIPTION:
The SARveillance trial is an efficient, pragmatic, multi-centre, international, stratified, partially-randomised, patient-preference trial within a registry of high versus lower intensity radiological surveillance following primary resection of retroperitoneal, abdominal and pelvic soft tissue sarcoma. The trial design is stratified by sarcoma tumour grade (high/intermediate grade and low grade). Both high and lower intensity follow-up represent current practice in different centres across the trial delivery network, with variation at a centre and surgeon level. SARveillance is co-produced in deep collaboration with a patient advisory group. The delivery network is trans-continental including major sarcoma centres in Europe, Asia, and the Americas with central coordination from Istituto Nazionale Tumori, Milan, Italy and Birmingham Centre for Observational and Prospective Studies (BiCOPS) University of Birmingham, UK. For centres that would otherwise be precluded from participating in SARveillance due to institutional level data sharing restrictions, provision has been made for prearranged Individual Participant Data Meta-Analysis (IPDMA). The IPDMA essentially replicates the instruments and processes of SARveillance at a single site level and allows for the PI to provide data for meta-analysis at the close of SARveillance, rather than sharing real-time data with the SARveillance servers at the coordinating institutions. Adult patients undergoing primary resection for retroperitoneal, abdominal and pelvic sarcoma will be eligible for inclusion. The trial design is innovative and efficient, implemented as a trial within an international registry, and adopting concepts from the pragmatic REaCT trial design methodology. Patients that are willing to be randomised will be allocated in a 1:1 ratio to a high or lower intensity follow-up schedule. For patients that decline randomisation, the trial has patient preference arms to maximise insight into decision-making processes in the context of a rare disease and maximise participant recruitment. The primary outcome measure is quality of life, measured as emotional functioning (EF) up to 5 years after surgery, measured 3-monthly, using the questions relating to the EF domain of the European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life questionnaire (QLQ-C30). Secondary outcomes for the trial will be overall survival up to 5 years after surgery, the cancer worry scale (EORTC library), health utility calculated using EuroQol Group EQ-5D-5L and cost-effectiveness health utility, measured using EQ-5D-5L. The primary outcome measure for low grade tumours is health utility. Pre-planned sub-studies will be conducted including an economic analysis, and validation study for a prognostic risk model.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 18 years)
* Primary resection
* Histologically confirmed retroperitoneal, abdominal or pelvic soft tissue sarcoma
* R0/R1 resection
* Eligible whether or not the participant undergoes neoadjuvant treatment

Exclusion Criteria:

* Metastatic disease at time of randomisation
* Recurrent, metastatic or residual disease identified on baseline CT imaging (3-4 months post primary resection)
* Reoperation for recurrent soft tissue sarcoma
* Re-resection following previous inadequate surgery
* R2 resection
* Patients receiving adjuvant therapy that will delay, interrupt or render radiological surveillance unpredictable
* Uterine sarcomas, gastrointestinal stromal tumour (GIST), fibromatosis, epithelial tumours, multifocal disease, sarcomas of bony origin
* Patient declined to consent to data sharing with RESAR (unless in a centre contributing via pre-planned IPDMA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Emotional Functioning | 5 years
  Quality of life, assessed using Emotional Functioning domain (items 21-24) of the European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life questionnaire (QLQ-C30). Each of the four items for this functional domain are scored between 1 and 4 (range: 3) to a total of 16 points, scaled to a total out of 100 using a validated formula from the EORTC scoring manual.

SECONDARY OUTCOMES:
Overall survival | 5 years
  From time of primary surgery to death (all-cause mortality) or last follow up
Cancer worry scale | 5 years
  Cancer-worry, assessed using four specific items from the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life item library. Each of the four items are scored between 1 and 4 (range: 3) to a total of 16 points, scaled to a total out of 100 using a validated formula from the EORTC scoring manual.
Health utility | 5 years
  EuroQol Group EQ-5D-5L. Each of the five items are scored between 1 and 5 (range: 4) to a total of 25 points, scaled to a weighted index between 0 and 1 using a validated formula from the EUROQOL scoring manual.

OTHER OUTCOMES:
Disease free survival | 5 years
  Defined as time from primary surgery to radiological evidence of disease recurrence as defined by the revised-RECIST criteria, by definition will be decreased in the high intensity follow-up group. This will be adopted as a process measure rather than an outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Ford, PhD, Principal Investigator — samuel.ford@uhb.nhs.uk
Locations (2):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy, Italy
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For international centres that would otherwise be precluded from participating in SARveillance, due to institutional level data sharing restrictions, provision has been made for prearranged Individual Participant Data Meta-Analysis (IPDMA). The IPDMA essentially replicates the instruments and processes of SARveillance at a single site level and allows for the PI to provide data for meta-analysis at the close of SARveillance. As the IPDMA derived data is supported by identical trial processes and materials, the subsequent data submitted for meta-analysis will be comparable in quality, safeguarding the statistical integrity of SARveillance during the meta-analysis. Centres within the trial delivery network that utilise the IPDMA process will be internal sponsors for SARveillance at the institutional level and are required to complete a pre-emptive agreement to share unidentified data with the trial network coordinating institutions for meta-analysis when SARveillance closes.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon locking the study database upon completion of last patient's follow-up.
Access Criteria: After approval by the central Trial Management group and completion of a study data sharing agreement.

REFERENCES:
- [Background] Baia M, Ford SJ, Dumitra S, Sama L, Naumann DN, Spolverato G, Callegaro D. Follow-up of patients with retroperitoneal sarcoma. Eur J Surg Oncol. 2023 Jun;49(6):1125-1132. doi: 10.1016/j.ejso.2022.02.016. Epub 2022 Mar 4. PMID 35277304
- See also: TARPSWG July 2020 - Trial development meeting — https://tarpswg.org/wp-content/uploads/2020/07/8.sarveillance-tarpswg-meeting-july-2020.pdf
- See also: RCSEd Pump Priming Grant funding — https://rcsed.shorthandstories.com/march-awards-grants/index.html